CLINICAL TRIAL: NCT05259137
Title: Intra-lesional ACE Inhibitor for Treatment of Hypertrophic Scars
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study never began, it did not proceed beyond an initial REB review
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24816
Record Dates: First submitted 2022-02-08; First posted 2022-02-28 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Hypertrophic Scar
Keywords: Keloid; Scar; Hypertrophy; ACE inhibitor; Angiotensin converting enzyme inhibitor; Enalapril; Hypertrophic
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid; Cicatrix; Hypertrophy | interventions — Enalaprilat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intra-lesional triamcinolone acetonide (No Intervention): This arm will will be our control. They will receive current standard of care of a single intra-lesional injection of 1 mL of 10mg/mL triamcinolone acetonide at 0 weeks, 6 weeks, and 12 weeks.
- Intra-lesional triamcinolone acetonide + enalaprilat (Experimental): This will be our intervention experiment. They will receive a single intra-lesional injection of 1.0 mL of 1.25 mg/mL of enalaprilat at 0 weeks, 6 weeks, and 12 weeks.
  Interventions: Drug: Intralesional enalaprilat injection

INTERVENTIONS:
Drug: Intralesional enalaprilat injection — 1.0 mL of 1.25 mg/mL enalaprilat
  Other Names: Enalaprilat
  Arms: Intra-lesional triamcinolone acetonide + enalaprilat

SUMMARY:
Hypertrophic scarring is a difficult and debilitating condition where one develops excessive scarring after full thickness injury to the skin. This is very common in full thickness burn injury. Currently, there is no reliable treatment of these scars. One of the more effective treatments available is serial intralesional injection of a steroid.

Angiotensin II is an active peptide in the body that results in vasoconstriction of the blood vessels when activated. Medications used today like angiotensin II receptor blocks and angiotensin converting enzyme inhibitors work to prevent the activation of angiotensin II and are mainly used to help control blood pressure. Previous studies in rat models have shown that angiotensin II receptor blockers can effectively reduce scar hypertrophy.

In this study, the investigators will conduct a randomized control trial with a paired split-scar design. One arm receiving the standard therapy of serial intra-lesional injections of triamcinolone acetonide (TAC) and the second arm receiving an ACE-inhibitor. The outcome will be measured using the Patient and Observer Scar Assessment Scale (POSAS), a validated assessment tool.

DETAILED DESCRIPTION:
Intralesional injection of corticosteroids such as triamcinolone acetonide (TAC) for treatment of hypertrophic scars are often used as first-line therapy owing to their ease of administration and relatively low cost. This medication mitigates further scar growth through increasing local vasoconstriction and simultaneously decreasing local inflammation at the site of scar hypertrophy.

Angiotensin II is an active peptide hormone which is produced by a cascade of reactions in order create its final form. Angiotensin converting enzyme (ACE) inhibitors, such as enalaprilat, competitively inhibit the enzyme that converts angiotensin I to angiotensin II. Angiotensin II receptor blockers, such as losartan, competitively inhibit the receptor. Both cause a decrease in the active form of angiotensin II and angiotensin II-induced vasoconstriction, resulting in lower blood pressure. Losartan has been demonstrated in rat models to effectively reduce the incidence of scar hypertrophy when administered post-operatively. With scar hypertrophy there is an overactivation of the wound healing cascade in both hypertrophic and keloid scars. As its vasodilative effects can be elicited without metabolism by the liver, local injection of either and ACE inhibitor or an ARB is hypothesized to effectively decrease the local effects of hypertrophy in scars.

Enalaprilat is an ACE-inhibitor that is used to treat hypertension and given in intravenous form. It is approved by Health Canada for this use. TAC is a synthetic glucocorticoid corticosteroid with marked anti-inflammatory action. It is approved by Health Canada. It is suitable for intradermal, intra-articular, and intrabursal injection.

In this study, the investigators plan to conduct a randomized control trial to determine the efficacy of intralesional injection of enalaprilat, an ACE-inhibitor, for treatment of hypertrophic scarring. Current standard of practice at the Halifax Infirmary consists of serial injections of TAC at the time of excision and then every 6 weeks for a total of three injections. The investigators plan to test this method against the injection of intralesional enalaprilat. The trial will be carried in compliance with the protocol, Canadian guidelines for Good Clinical Practice and the research ethics board of Nova Scotia Health Authority.

The investigators propose a double-blinded randomized controlled trial with a paired split-scar design to test the use of enalaprilat for intralesional injection in a hypertrophic scar. This will be compared against injection of TAC alone, the standard of care for hypertrophic scarring. The objective of this trial is improvement in the hypertrophic scar with the use of enalaprilat as measured by the Patient and Observer Scar Assessment Scale.

This study will be a randomized, double-blind, human clinical trial. In compliance with the CONSORT (Consolidated Standards of Reporting Trials) guidelines, this trial will be registered with the International Standard Randomized Controlled Trial Number registry.

Participants will be recruited from the Health Infirmary plastic surgery outpatient clinics in Halifax, Nova Scotia, Canada. Inclusion criteria will be: Patients with scar tissue demonstrating features of hypertrophic scarring (e.g., raised, red tissue, contractures) Clinical office will be the site of intra-lesional injection as conditions are optimal with consistent lighting, tools/equipment, and support personnel. Exclusion criteria will be: (1) scar does not demonstrate any distinguishing features of hypertrophic scar; (2) self-reported as pregnant and/or breastfeeding; (3) documented hepatic, heart, or renal dysfunction; (4) patients with known Cushing's disease or glaucoma; (5) documented history of angioedema; (6) patients with diabetes; (7) patients being treated with any anti-hypertensive medications (8) patients under 18 years of age. Once patients have been identified the nature of the study will be explained and consent will be obtained verbally and in writing for treatment and involvement in the study. The following variables will be extracted from each participant: (1) age, (2) gender, (3) smoking status, and (4) comorbidities.

Patients will receive both arms of treatment as per the split scar study design. In order to ensure that there is limited chance for breaking treatment codes, a Microsoft excel sheet will be used to keep track of assigned participants and held by a third party with no involvement with the trial. Should a patient develop an adverse event to the treatment, the third party will break code and reveal only their assigned group. The patient in question will then be removed from the study to ensure confidentiality.

Once patients have been identified with a hypertrophic scar and consented, they will undergo pre-operative baseline assessments. The POSAS will be used to rate a baseline evaluation of the participant's scar. On this initial evaluation participants will be stratified into mild, moderate, and severe hypertrophic scarring, and randomisation will occur within each stratum using their study identifier assigned by study staff. Patients will then be administered an intralesional injection of either 1 mL of enalaprilat [1.25 mg/mL] (intervention group) or 1 mL TAC [10 mg/mL] (control group) under the care of attending plastic surgeon.

Enalaprilat and TAC are non-toxic substance commonly found in the hospital setting and disposed of using no precautions, therefore no accountability procedures are necessary for the use of these substances for the duration of the clinical trial. All rescue medications used to treat the unlikely event of an allergic reaction are permitted. There are no antidotes available for the use of enalaprilat.

Postoperative follow-up will be completed at the Halifax Health Infirmary. The primary endpoint will be resolution of the hypertrophic scar or improvement of the hypertrophic scar assessed using the POSAS evaluations. The secondary endpoint will be recurrence, worsening, or failure of improvement of their hypertrophic scar. POSAS evaluations conducted by blinded participants (for patient-reported POSAS) and blinded study staff evaluators (for observer-reported POSAS) will be completed at 6-, 12-, and 52 weeks post-injection in the general plastic surgery clinic in the Halifax Infirmary. General assessment of participant health status and wellbeing will be completed during the same follow-up visits to track other adverse reactions to treatments. Patients will also have access to the plastic surgery on-call service should they have any concerns.

Discontinuation of the trial will happen if recurrence of hypertrophic scarring is significantly higher (p<0.05) than the control.

Patients are able to withdraw at any point with no consequences. Should a patient withdraw all of their information up to the timing of withdrawal, excluding demographic information, will be removed from the study. Patients who withdraw will be replaced in a randomized fashion in order to ensure suitable numbers of CN and EX groups. Patients who withdraw will be followed up by their respective plastic surgeon as would be customary for treatment of hypertrophic scarring.

All trial patients will be monitored at each contact with a healthcare professional during the trial for potential adverse events. This will happen at 0, 6, 12, and 52 weeks as per the study design. Patients will also be able to schedule appointments outside of the normal follow-up. They will be assessed at these times. Plastic surgeons and study evaluators will notify the principal investigator should an adverse event occur. The principal investigator will then report to Health Canada using the Adverse Drug Reactions form immediately. Patients who develop an adverse drug reaction will be followed up bi-weekly by their attending plastic surgeon until cessation of symptoms for one month.

Each individual parameter included in the POSAS, as well as the overall scores, will be analyzed using an ANOVA. Comparisons will be made within each stratum (mild, moderate, or severe) in order to identify the effect of the treatment alone without respect to the severity of the scar evaluated at baseline. Comparisons will also be made between strata in order to determine if efficacy levels of each treatment with respect to baseline severity of the scar.

Due to the lack of effect size data reported on this administration route for enalaprilat, a formal power analysis cannot be provided. This study poses as an exploratory investigation into the efficacy of enalaprilat in the treatment of hypertrophic scars in response to findings using losartan in rat models that demonstrated its effective use in the reduction of hypertrophy incidence when administered post-operatively. For this reason, 30 participants was determined to be sufficient.

POSAS results will be collected directly onto physical copies of the POSAS v2.0. Treatment dosages will be recorded on clinic visit files and transferred to a de-identified study file linked to participant study identifiers for documentation.

All demographic records, POSAS evaluations, and any other data pertaining to study participants will be managed by the Primary Investigator and research coordinator. Data will be de-identified by one of these two individuals before becoming accessible by all study staff and provided to the Division of Plastic Surgery. A file of data aligning participant identities to study identifiers will be maintained by the Principal Investigator.

De-identified trial data will be available only to assigned trial personnel identified in this application. Participants will not be identified in any way in reports or publications as a result of participation in this trial. All de-identified trial data will be kept for 25 years per Halifax Infirmary requirements. Only data required by any scientific journals, regulatory agencies, or applicable organisations will be kept beyond 25 years.

ARBs and ACE inhibitors have been used subcutaneously safely in investigations of its systemic effects. Failure of enalarilat to effectively reduce the hypertrophic scar is equivalent to no treatment on the scar and therefore, participants who respond unfavorably to interventional injection will be given the option to complete a full course of control treatment at the end of their follow-up evaluation schedule. In order to mitigate risk in the unexpected event of an allergic and/or anaphylactic reaction, participants will be briefly monitored after enalaprilat injection.

Research Ethics Board (REB) Review and Informed Consent i. Informed consent is to be obtained as per the institutional SOP for Requirements (701) and Documentation (703) of Informed Consent.

iii. Effects of study-related bias is minimised by the randomised assignment of participants in control or interventional study groups. Participant patients will be handled under the care of Supervising Investigator, Dr Michael Bezuhly, in the general plastic surgery clinic at the Halifax Infirmary. Eligible participants are determined on the day of the injection after their study group has been assigned.

iv. Conflicts of interest: Participant patients will be handled under the care of Supervising Investigator, Dr Michael Bezuhly, in the general plastic surgery clinic at the Halifax Infirmary. Dr Bezuhly has no disclosures.

Participant Confidentiality All demographic records, POSAS evaluations, and any other data pertaining to study participants will be entirely confidential. Assessing and comparing the interventions underwent in this study does not require data to be linked to specific patients. If a participant chooses to withdraw from the study or in the case of an audit, participant data will be de-identified using that participant's study identifier. A file of this data aligning participant identities to study identifiers will be maintained by the Principal Investigator.

De-identified trial data will be available only to assigned trial personnel identified in this application. Participants will not be identified in any way in reports or publications as a result of participation in this trial. All de-identified trial data will be kept for 25 years per the Halifax Infirmary requirements.

Study Modification and Discontinuation Study participants may withdraw their consent and inclusion in the study at any time. Further data for these participants will not be collected and their existing information will be excluded from further the data analyses. The Halifax Infirmary Research Ethics Board and the principal investigator retain the right to terminate patient recruitment or cancel the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with scar tissue demonstrating features of hypertrophic scarring (e.g., raised, red tissue, contractures, extends beyond the boundary of the original wound)

Exclusion Criteria:

1. scar does not demonstrate any distinguishing features of hypertrophic scar;
2. self-reported as pregnant and/or breastfeeding;
3. documented hepatic, heart, or renal dysfunction;
4. patients with known Cushing's disease or glaucoma;
5. documented history of angioedema;
6. patients with diabetes;
7. patients being treated with any anti-hypertensive medications
8. patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Patient and Observer Scar Assessment Scale (POSAS) | Outcomes will be measured at 0, 6-, 12-, and 52 weeks
  The POSAS patient scale uses patient-reported measurements of symptoms (pain and itchiness) and signs (colour, stiffness, thickness, irregularity) to quantify the degree of the scar. Similarly, the POSAS observer scale uses measurements of scar vascularity, pigmentation, thickness, relief, pliability, and surface area in order to quantify development of scar tissue. For the observer, the maximum score is 50 and the minimum score is 5. A higher score indicates a worse outcome. For the patient, the maximum score is 60 and the minimum score is 6. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bezuhly, MD, MSc, Study Director — Dalhousie University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barone N, Safran T, Vorstenbosch J, Davison PG, Cugno S, Murphy AM. Current Advances in Hypertrophic Scar and Keloid Management. Semin Plast Surg. 2021 Aug;35(3):145-152. doi: 10.1055/s-0041-1731461. Epub 2021 Jul 15. PMID 34526861
- [Background] Kaschina E, Unger T. Angiotensin AT1/AT2 receptors: regulation, signalling and function. Blood Press. 2003;12(2):70-88. doi: 10.1080/08037050310001057. PMID 12797627
- [Background] Griffith BH. The treatment of keloids with triamcinolone acetonide. Plast Reconstr Surg. 1966 Sep;38(3):202-8. doi: 10.1097/00006534-196609000-00004. No abstract available. PMID 5919603
- [Background] Al-Attar A, Mess S, Thomassen JM, Kauffman CL, Davison SP. Keloid pathogenesis and treatment. Plast Reconstr Surg. 2006 Jan;117(1):286-300. doi: 10.1097/01.prs.0000195073.73580.46. PMID 16404281
- [Background] Niessen FB, Spauwen PH, Schalkwijk J, Kon M. On the nature of hypertrophic scars and keloids: a review. Plast Reconstr Surg. 1999 Oct;104(5):1435-58. doi: 10.1097/00006534-199910000-00031. No abstract available. PMID 10513931
- [Background] Chatterjee K, De Marco T. Systemic and coronary haemodynamics and pharmacodynamics of enalapril and enalaprilat in congestive heart failure. Drugs. 1990;39 Suppl 4:29-40; discussion 41-2. doi: 10.2165/00003495-199000394-00007. PMID 2162294
- [Background] Franchignoni F, Giordano A, Vercelli S, Bravini E, Stissi V, Ferriero G. Rasch Analysis of the Patient and Observer Scar Assessment Scale in Linear Scars: Suggestions for a Patient and Observer Scar Assessment Scale v2.1. Plast Reconstr Surg. 2019 Dec;144(6):1073e-1079e. doi: 10.1097/PRS.0000000000006265. PMID 31764669
- [Background] Danielsen PL, Rea SM, Wood FM, Fear MW, Viola HM, Hool LC, Gankande TU, Alghamdi M, Stevenson AW, Manzur M, Wallace HJ. Verapamil is Less Effective than Triamcinolone for Prevention of Keloid Scar Recurrence After Excision in a Randomized Controlled Trial. Acta Derm Venereol. 2016 Aug 23;96(6):774-8. doi: 10.2340/00015555-2384. PMID 26911400
- [Result] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Result] Juckett G, Hartman-Adams H. Management of keloids and hypertrophic scars. Am Fam Physician. 2009 Aug 1;80(3):253-60. PMID 19621835
- [Result] Kawano Y, Yoshida K, Matsuoka H, Omae T. Chronic effects of central and systemic administration of losartan on blood pressure and baroreceptor reflex in spontaneously hypertensive rats. Am J Hypertens. 1994 Jun;7(6):536-42. doi: 10.1093/ajh/7.6.536. PMID 7917152
- [Result] Morelli Coppola M, Salzillo R, Segreto F, Persichetti P. Triamcinolone acetonide intralesional injection for the treatment of keloid scars: patient selection and perspectives. Clin Cosmet Investig Dermatol. 2018 Jul 24;11:387-396. doi: 10.2147/CCID.S133672. eCollection 2018. PMID 30087573
- [Result] Murphy A, LeVatte T, Boudreau C, Midgen C, Gratzer P, Marshall J, Bezuhly M. Angiotensin II Type I Receptor Blockade Is Associated with Decreased Cutaneous Scar Formation in a Rat Model. Plast Reconstr Surg. 2019 Nov;144(5):803e-813e. doi: 10.1097/PRS.0000000000006173. PMID 31385893
- [Result] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683